CLINICAL TRIAL: NCT06318910
Title: Effects of Customized Foot Orthoses With Orthotic Wedges on Lower-extremity Muscle Activity During Standing and Gait in the Patients With Plantar Heel Pain: A Randomized Controlled Trial
Brief Title: Customized Foot Orthoses on Muscle Activity During Standing and Gait in Plantar Heel Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MU-SRF-RS-27 C/66
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Foot Orthoses; Fasciitis, Plantar
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: The present study will use a randomized controlled trial (RCT) to determine the effectiveness of CFO for the treatment of patients with PHP. Three treatment groups including the CFO without wedge, the CFO with W1, and the CFO with W2 will be randomly assigned to each participant by a computer-generated randomization. The opaque-sealed envelopes will be used to allocate the groups of participant.
Who Masked: Outcomes Assessor
Masking Description: Participants will be allocated to the control (CFO without wedge) or experimental (CFO with W1 or W2) groups according to the seal-envelop randomization technique. Then, they will be assessed all outcomes for the baseline including pain intensity, foot function, lower-extremity muscle activity during gait and standing by the 2nd physical therapist. And the participants will receive the assigned treatment by the 1st physical therapist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CFO with W1 (Experimental): The therapists will propose the orthotic wedges after examining the foot angles following the foot assessment from the study of Root, the forefoot angle will be determined for both the forefoot and rearfoot wedges. Previous studies recommended the posting at 60% of the measured forefoot angle, up to a maximum of 8 degrees, for extrinsic forefoot varus wedge and the posting at 50% of the measured forefoot angle, up to a maximum of 6 degrees, for extrinsic rearfoot varus wedge. After the posting, all participants will be asked to test the provided foot orthoses within their footwear. If any disturbance has been found during testing, the adjustment will be performed.
  Interventions: Device: orthotic wedge; Device: CFO
- CFO with W2 (Experimental): The therapists will propose the orthotic wedges after examining the foot angles following the foot assessment from the study of Monaghan et al., the forefoot will be posted at 50% of the measured forefoot angle, and the rearfoot will be posted at 20% of the measured rearfoot angle. After the posting, all participants will be asked to test the provided foot orthoses within their footwear. If any disturbance has been found during testing, the adjustment will be performed.
  Interventions: Device: orthotic wedge; Device: CFO
- CFO without wedge (Active Comparator): The 3-quarter-length CFO will be made from thermoplastic material (rigid foot orthoses) which consists of four layers i.e. two layers of 0.5-mm polyvinyl chloride (PVC), one layer of 1.5-mm thick fiber to increase strength of foot orthoses in the bottom layers as well as one layer of 1.2-mm genuine leather in the upper layer to increase comfort. It incorporates a heat-molding process to adjust individual foot shape in prone position. The materials will be set within approximately three minutes.
  Interventions: Device: CFO

INTERVENTIONS:
Device: orthotic wedge — The orthotic wedges with a full length of 3-mm soft foam layer will be provided to each participant under the molded orthoses; the amount of wedge angle will depend on the rearfoot and forefoot angles of the participants. The present study developed 3-degree, 6-degree, and 8-degree wedges for the rearfoot and forefoot. It was made from solid rubber with a cover of thin fabric. There are three sizes for these products which include small (S), medium (M), and large (L) sizes, according to the foot length of participants.
  Arms: CFO with W1; CFO with W2
Device: CFO — The 3-quarter-length CFO will be made from thermoplastic material (rigid foot orthoses) which consists of four layers i.e. two layers of 0.5-mm polyvinyl chloride (PVC), one layer of 1.5-mm thick fiber to increase strength of foot orthoses in the bottom layers as well as one layer of 1.2-mm genuine leather in the upper layer to increase comfort. It incorporates a heat-molding process to adjust individual foot shape in prone position. The materials will be set within approximately three minutes.

SUMMARY:
The present study will use a randomized controlled trial (RCT) to determine the effectiveness of customized foot orthosis (CFO) for the treatment of patients with PHP. Three treatment groups including the CFO without wedge, the CFO with wedge type 1 (W1), and the CFO with wedge type 2 (W2) will be randomly assigned to each participant by a computer-generated randomization. The opaque-sealed envelopes will be used to allocate the groups of participant.

DETAILED DESCRIPTION:
Participants will be allocated to the control (CFO without wedge) or experimental (CFO with W1 or W2) groups according to the seal-envelop randomization technique. Then, they will be assessed all outcomes for the baseline including pain intensity, foot function, lower-extremity muscle activity during gait and standing by the 2nd physical therapist. And the participants will receive the assigned treatment by the 1st physical therapist.

All participants will be asked to use the CFO in daily life during weight-bearing activities, and logbook, chat LINE, or phone call will be used to monitor the participants during the treatment program. They will be asked about activity they done in daily and a number of hour they used CFO per day in diary book. At least 4 hours per day of wearing CFO will be required to each participant. After 3 months of the CFO use, all outcomes will be re-assessed by the 2nd physical therapist. And such outcomes will be then statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Reaching the specific criteria of PHP including

  * A complaint of tenderness from the palpation of the medial calcaneal tubercle and the medial aspect of the proximal portion of the plantar fascia, or pain along the plantar fascia at medial longitudinal arch side
  * The presence of heel pain immediately during the first few steps of walking in the morning or after a prolonged period of inactivity; and gradually decreased throughout the day with ordinary walking, and worsened with prolonged activity
* Having the symptom of heel pain for at least 6 weeks, indicates the chronic condition
* Having the maximum level of pain intensity during last week using the visual analog scale (VAS) at least 3 out of a full 10 scores

Exclusion Criteria:

* Having positive sciatica test, indicating the L5-S1 nerve root irritation
* Having a history of lower extremity fracture
* Having a history of lower extremity surgery
* Having been diagnosed with gout, diabetic neuropathy, rheumatoid arthritis, systemic lupus erythematosus (SLE), cancer, infectious disease, and tumor

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity and foot function | Baseline, 3 months
  Pain intensity during the last week will be assessed using the visual analog scale (VAS) which is the high-reliability measurement (ICC = 0.88). The highest pain level is 10 and the lowest pain level is 0. In addition, the foot function will be assessed by the 23-item foot function index (FFI). The present study will use the Thai version of FFI that has been translated forward and backward from the English version. The previous study showed high internal consistency (Cronbach alpha = 0.98) and high test-retest reliability (ICC = 0.86). It is appropriate to use among patients with PHP.
EMG of lower leg muscles | Baseline, 3 months
  A Trigno Wireless EMG system at 2000 Hz (Delsys Inc., Boston, MA) will be used to collect the EMG data from Tibialis anterior, Peroneus longus, Medial gastrocnemius, Biceps femoris, and Rectus femoris in both legs. The skin will be cleaned with alcohol wipes and the standard EMG electrodes will be positioned following the SENIAM guidelines. Raw EMG data will be exported to Visual3D (C-Motion Inc., Germantown, USA). The dependent variables for the peak and integrated EMG (iEMG) values from such muscles will be found. Then, the data will be normalized to the maximal observed signal during the dynamic contraction during the movement tasks. The participants will be asked to stand with both legs on the firm and foam surface in two conditions i.e. eye closed and eye open, for 20 s in each condition. And then, they will be asked to walk at a self-selected speed to the other end of the 3-m pressure distribution platform.

OTHER OUTCOMES:
Subjective assessment | Baseline
  A self-reported questionnaire will be divided into 4 parts, including individual information (i.e. sex, age, gender, dominant side, body mass index, job, average time during standing and walking), general health information (i.e. characteristics of heel pain, history of injury and fracture at the lower extremity, falling history, types of footwear), foot pain and function, low back pain and lower-extremity pain.
Physical assessment | Baseline
  Physical characteristics of the participants will be assessed by the 1st physical therapist, including measurements of standing posture, leg length, quadriceps angle, tibiofemoral angle, knee recurvatum, dorsiflexion lunge test, navicular drop test, first metatarsophalangeal joint angle and posture, foot posture during standing and prone lying, neural tension test, lateral step down test, and star excursion balance test. Intra-rater reliability from data of each physical assessment among 10 persons showed the Intraclass Correlation Coefficients ICC(3,1) values ranging from 0.69 to 0.98.